CLINICAL TRIAL: NCT06217913
Title: Effects of Monitoring Blood Pressure in High-risk Pregnant Women Using a Wearable Device
Brief Title: Effects of Monitoring Blood Pressure During Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: XH-23-010
Record Dates: First submitted 2023-08-25; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-08

CONDITIONS: Birth Weight; Weight Gain Trajectory
MeSH Terms: conditions — Birth Weight; Body-Weight Trajectory

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): routine delivery examination group
- intervention group (Experimental): routine delivery examination group + use of wearable blood pressure monitoring device group
  Interventions: Device: wearable device to monitor the blood pressure

INTERVENTIONS:
Device: wearable device to monitor the blood pressure — Pregnant women began to establish antenatal examination records (usually before 12 weeks of pregnancy), and were enrolled through randomized grouping. Pregnant women in the intervention group were provided with wearable blood pressure monitoring equipment, and ambulate blood pressure monitoring was conducted for at least 2 24 hours per week from 12 weeks of pregnancy until 28 weeks of pregnancy, after which blood pressure monitoring was carried out according to routine antenatal examination.
  Arms: intervention group

SUMMARY:
In this study, at least 400 women with high-risk of pregnancy hypertension will use a wearable device to monitor the blood pressure during gestational age from 12 weeks to 28weeks. The observed outcomes including maternal and offspring. Participants were from three hospital including Shanghai Xinhua Hospital, Jiaxing Maternal and Child Health Hospital and Peking University Third Hospital. Pregnant women were randomly divided into control group (routine delivery examination group) and intervention group (routine delivery examination group + use of wearable blood pressure monitoring device group), 200 cases each.

ELIGIBILITY:
Inclusion Criteria:

* Women with a single pregnancy before 12 weeks of pregnancy
* The presence of any of the following risk factors: age > 30 years, a history of eclampsia, a family history of eclampsia, obesity (BMI ≥ 30 Kg/m2), and a history of gestational hyperglycemia (pregestational type 1 and type 2 diabetes; gestational manifest diabetes and gestational diabetes requiring insulin treatment), preexisting chronic hypertension, kidney disease, and autoimmune diseases such as systemic lupus erythematosus and antiphospholipid syndrome.
* Signed the informed consent can be continuously followed up.
* Permanent population living in the study area.
* All subjects received routine antenatal examination and treatment.

Exclusion Criteria:

* Termination of pregnancy before 20 weeks
* Withdraw from the study
* Lost visitors

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Offspring weight change | up to 24 months
  The offspring would be followed up from birth to 2 years of age at 42days, 3, 6, 12, 18 and 24 months of birth. Birth weights and weights would be measure in kilograms. The primary outcome the growth curve of the follow-up weights.

SECONDARY OUTCOMES:
Maternal blood pressure change | 16 weeks
  24-hour weekly blood pressure and its fluctuation in pregnant women from 12 to 20 weeks of gestation would be measure in mmHg.
Maternal complications | 28 weeks
  The incidence of hypertension in pregnancy, pre-eclampsia, eclampsia, placental abruption, transient ischemic attack or stroke, and HELLP syndrome, which would be stated in percentages.
Offspring outcomes | up to 24 months
  Including incidence such as neonatal respiratory distress syndrome, sepsis, early-onset thrombocytopenia, early-onset neutropenia, hypoglycemia, congenital hypothyroidism, bronchopulmonary dysplasia, necrotizing enterocolitis, recurrent respiratory infections, infantile wheeze etc., which would be stated in percentages.
Offspring neurodevelopment | up to 24 months
  Assessing neurodevelopment using ASQ scores or Bayley scores.
Offspring perinatal outcomes | up to 24 months
  Including the incidence of mortality, large for large for gestational age infants and small for gestational age infants, which would be stated in percentages.

OTHER OUTCOMES:
metabolomics | 16 weeks
  Meteranl metabolomics during pregnancy (around gestational age at 12 weeks and 28weeks) would be measured in pg/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No